CLINICAL TRIAL: NCT05130307
Title: Virtual Reality Analgesia for Brief Thermal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Hunter Hoffman, Affiliate Assistant Professor, Psychology, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00013916
Record Dates: First submitted 2021-11-01; First posted 2021-11-23 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Pain, Acute
Keywords: Pain control
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: A Mixed Model repeated measures ANOVA or non-parametric tests if appropriate will be conducted on worst pain ratings. Within subjects crossover design, VR treatment order randomized (some participants receive order 1 Low Tech VR + High Tech VR = Arm 1, some participants receive order 2 High Tech VR + Low Tech VR) = Arm 2.
  . Treatment order 1: Low Tech/less interactive Virtual Reality for 1st brief pain stimulus+ washout period + High Tech for 2nd brief pain stimulus.
  Treatment order 2: High Tech/more interactive VR for 1st brief pain stimulus + washout period + Low Tech for 2nd brief pain stimulus (Arm 2)..
Who Masked: Participant
Masking Description: Although no deception is involved, participants who receive VR will remain unaware of the immersiveness of the VR systems they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Order 1 (Experimental): Treatment order 1: Low Tech (less interactive) Virtual Reality for 1st pain stimulus+ High Tech for 2nd pain stimulus
  Interventions: Behavioral: virtual reality game
- Treatment Order 2 (Active Comparator): Treatment order 2: High Tech VR (more interactive) for 1st pain stimulus + Low Tech for 2nd pain stimulus.
  Interventions: Behavioral: virtual reality game

INTERVENTIONS:
Behavioral: virtual reality game — participants interact with a computer generated world

SUMMARY:
Using immersive virtual reality as a form of pain distraction during a brief "painful but tolerable" temperature.

DETAILED DESCRIPTION:
This study will use Quantitative Sensory Testing (computer-controlled brief 10 second thermal pain stimuli) in healthy college students.

The primary aim is to conduct a randomized, controlled study with healthy volunteers to explore whether interacting with virtual objects in VR via a highly immersive VR system makes VR significantly more effective/powerful compared to a less immersive VR system, vs. No VR, for reducing pain during quantitative sensory testing.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a course at the University of Washington Psychology Dept., participating in the UW Psychology subject pool
* Able to read, write and comprehend English
* Able to complete study measures
* Willing to follow our UW approved instructions
* 18 years of age or older
* Currently enrolled in a course at the University of Washington Psychology Dept., participating in the UW Psychology subject pool
* Able to read, write and comprehend English
* Able to complete study measures
* Willing to follow our UW approved instructions
* 18 years of age or older The following temporary inclusion/exclusion criterion will exist only as long as required or appropriate for COVID pandemic conditions.

COVID-19 precautions. Vaccinated: Individuals are considered fully vaccinated 2 weeks after the second dose in a 2-dose series (e.g., Pfizer or Moderna) or 2 weeks after a single-dose vaccine (e.g., Johnson & Johnson).

All students and researchers must wear masks at all times during the study, and participants and researchers must provide proof of full vaccination for full participation.

If participants do not have proof of vaccination or are unvaccinated, they are still free to sign up for the study. They are invited. They can still earn the extra credit by reading educational materials, in person, during their scheduled time slot. If unvaccinated, or if they have no proof of vaccination, we request that students provide proof of a negative COVID-19 test from the UW test site at the faculty lounge, dated within 24 hours of the study (non-vaccinated students need a recent negative COVID-19 test from the UW before participating in the non-VR educational materials option.

-

Exclusion Criteria:

* People how have already previously participated in this same study (e.g., last quarter) are not eligible to participate again.
* Not enrolled in a course at the University of Washington Psychology Dept., participating in the UW Psychology subject pool
* Not be able to read, write and comprehend English
* Younger than 18 years of age.
* Not capable of completing measures
* Not capable of indicating pain intensity,
* Not capable of filling out study measures,
* Extreme susceptibility to motion sickness,
* Seizure history,
* Unusual sensitivity or lack of sensitivity to pain,
* Sensitive skin,
* Sensitive feet
* Migraines
* Diabetes

The following temporary inclusion/exclusion criterion will exist only as long as required or appropriate for COVID pandemic conditions.

COVID-19 precautions. Vaccinated: Individuals are considered fully vaccinated 2 weeks after the second dose in a 2-dose series (e.g., Pfizer or Moderna) or 2 weeks after a single-dose vaccine (e.g., Johnson & Johnson).

All students and researchers must wear masks at all times during the study, and participants and researchers must provide proof of full vaccination for full participation.

If participants do not have proof of vaccination or are unvaccinated, they are still free to sign up for the study. They are invited. They can still earn the extra credit by reading educational materials, in person, during their scheduled time slot. If unvaccinated, or if they have no proof of vaccination, we request that students provide proof of a negative COVID-19 test from the UW test site at the faculty lounge, dated within 24 hours of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Worst pain, baseline, participant's rating of "worst pain" during baseline measure | Immediately after a single 10 second test (no more than 10 minutes before the subsequent test stiim)
  Baseline, Worst pain rating using a single graphic rating scale, 0 = no pain, 10 = excruciating pain
participant's rating of "worst pain" during test phase | Immediately after each single 10 second test stimulus (< 10 minutes after baseline pain rating)
  Test phase, Worst pain rating using a single graphic rating scale, 0 = no pain, 10 = excruciating pain

SECONDARY OUTCOMES:
Baseline, participants rating of "time spent thinking about pain" | Immediately after a single 10 second test (no more than 10 minutes before the subsequent test stiim)
  Baseline Time thinking, Single a single graphic rating scale, 0 = none of the time, 10 = all of the time
Test Phase, participants rating of "time spent thinking about pain" during test phase | Immediately after each single 10 second test stimulus (< 10 minutes after baseline pain rating)
  Test phase, Time rating, using a single graphic rating scale, 0 = none of the time, 10 = all of the time
Baseline, participants rating of "pain unpleasantness" | Immediately after a single 10 second test (no more than 10 minutes before the subsequent test stiim)
  Baseline, Unpleasant rating, using single graphic rating scale, 0 = not unpleasant at all, 10 = excruciatingly unpleasant
Test phase, participants rating of "pain unpleasantness" during test phase | Immediately after each single 10 second test stimulus (< 10 minutes after baseline pain rating)
  Test phase, pain unpleasantness, 0 = not unpleasant at all, 10 = excruciatingly unpleasant
Baseline, participants rating of "Fun" during baseline | Immediately after a single 10 second test (no more than 10 minutes before the subsequent test stiim)
  Baseline fun, 0 = no fun at all, 10 = extremely fun
Test Phase, participants ratings of "Fun" during test phase | Immediately after each single 10 second test stimulus (< 10 minutes after baseline fun rating)
  Test phase fun, 0 = no fun at all, 10 = extremely fun
Baseline pain intensity: participants ratings of pain intensity during brief pair of 10 sec stimuli | Immediately after a single 10 second test (no more than 10 minutes before the subsequent test stiim)
  Baseline, pain intensity rating using a single graphic rating scale, 0 = no pain, 10 = excruciating pain
Accuracy on the odd number task during No VR, Low tech VR and High tech VR | No pain during this measure, measured within 10 minutes after the QST measures are completed.
  participants accuracy on the attention demanding "odd number" task (Hoffman, 2021)

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Hoffman, M.S., Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington (only Psych students eligible, public not eligible for participation), Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregated data will be provided upon request on a case by case basis (e.g., for meta-analyses).
Time Frame: any time after publication
Access Criteria: meta-analysis

REFERENCES:
- [Background] Al-Ghamdi NA, Meyer WJ 3rd, Atzori B, Alhalabi W, Seibel CC, Ullman D, Hoffman HG. Virtual Reality Analgesia With Interactive Eye Tracking During Brief Thermal Pain Stimuli: A Randomized Controlled Trial (Crossover Design). Front Hum Neurosci. 2020 Jan 23;13:467. doi: 10.3389/fnhum.2019.00467. eCollection 2019. PMID 32038200
- [Background] Hoffman HG. Interacting with virtual objects via embodied avatar hands reduces pain intensity and diverts attention. Sci Rep. 2021 May 21;11(1):10672. doi: 10.1038/s41598-021-89526-4. PMID 34021173